CLINICAL TRIAL: NCT00279708
Title: Atorvastatin as a Disease Modifying Agent in Stage II and III Pulmonary Sarcoidosis: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Atorvastatin to Treat Pulmonary Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joseph R. Fontana, M.D., Staff Clinician, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060072; 06-H-0072 (Other: NIH NHLBI)
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: Granulomatous Inflammation; Steroid-Sparing; Pulmonary Function; Sarcoidosis, Pulmonary; Statins (Atorvastatin); Biomarkers; Nitric Oxide; Disease Activity; Quality of Life; Corticosteroids; Pulmonary Sarcoidosis; Sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Atorvastatin) (Active Comparator): Atorvastatin: Subjects were assigned to the treatment intervention by way of double blind masking. Atorvastatin 80 mg/day was the initial treatment given, as tolerated for a 12 month period. During the study, a 50% dose reduction was applied for subjects meeting pre-specified criteria.
  Interventions: Drug: Atorvastatin
- Control Arm (Placebo) (Placebo Comparator): Placebo: In a double-blind fashion, subjects were assigned to receive the sham intervention which appeared the same as the intervention agent. For subjects meeting pre-specified criteria, a 50% dose reduction was applied during the 12 month treatment phase of the study: Placebo vs. Atorvastatin
  Interventions: Other: Placebo Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin — Placebo vs. Atorvastatin
  Other Names: Lipitor
  Arms: Intervention Arm (Atorvastatin)
Other: Placebo Oral Tablet — Placebo: Sham Therapy in an oral tablet formulation
  Other Names: Placebo
  Arms: Control Arm (Placebo)

SUMMARY:
This study will determine if atorvastatin (Lipitor) can help patients with pulmonary (lung) sarcoidosis and replace or reduce the need for patients to take steroids, such as prednisone. Sarcoidosis is an inflammatory disease that can affect nearly any part of the body. Pulmonary sarcoidosis may resolve on its own or it may progress to irreversible lung damage, disability, and death. Many sarcoidosis patients are treated with prednisone, but the drug is not effective in all patients, and it can cause serious side effects, such as high blood pressure, sugar diabetes, eye cataracts, and bone thinning.

Patients with stage II or III pulmonary sarcoidosis between 18 and 70 years of age who require prednisone may be eligible for this study. Candidates are screened with the tests and procedures described below.

Participants are randomly assigned to one of two treatment groups: one group takes atorvastatin; the other takes a placebo (a look-alike pill that has no active ingredient to fight sarcoidosis). Both groups take the pills by mouth once a day for 12 months. When treatment begins, participants begin to have their prednisone dosage tapered (reduced). The tapering is done over 8 weeks until the dose is reduced by 90 percent. Patients are evaluated periodically to determine if the two groups differ in how long they can remain on the reduced dose of prednisone without having their symptoms recur, requiring an increase in the prednisone dose. A full battery of tests is done at the initial screening visit and at the 26- and 52-week follow-up visits, requiring hospitalization for 3-5 days. Additional interim outpatient assessments are done at 6, 12, 18 and 36 weeks.

The full battery of tests at the initial screening and the 26- and 52-week visits includes the following:

* Medical history, physical examination, blood and urine tests, assessment of disease severity and activity.
* Questionnaires.
* Chest x-ray (CXR) and computed tomography (CT) scan.
* Abdominal ultrasound.
* Six-minute walk test (6MWT)
* Exercise testing and blood gases
* Pulmonary function tests (PFT)
* Maximum incremental ventilatory performance test (MIVP)
* Exhaled nitric oxide and carbon monoxide (Exhaled NO and CO)
* Bronchoscopy and lavage

Interim testing at 6, 12, 18 and 36 weeks includes PFT, MIVP, Exhaled NO and CO, CXR, questionnaire, blood tests, and 6MWT.

Six months after completing the study, participants fill out a questionnaire.

DETAILED DESCRIPTION:
Background

Sarcoidosis is a multi-system granulomatous inflammatory disease. Pulmonary involvement is most common. Patients typically experience fatigue, weakness and dyspnea. Respiratory muscle weakness, which may be secondary to granulomatous inflammation, is associated with dyspnea and decreased quality of life (QOL). The disease can remit spontaneously or become chronic, with exacerbations and remissions. In some patients, it can progress to pulmonary fibrosis and death. Granulomatous inflammation is characterized primarily by accumulation of monocytes, macrophages and activated T-lymphocytes, with increased production of key inflammatory mediators, TNF-alpha, INF-gamma, IL-2 and IL-12, characteristic of a Th1-polarized response (T-helper lymphocyte-1 response). Corticosteroids are the current mainstay of treatment, but their long-term benefits are not certain. Because steroids often produce undesirable side effects, investigations to identify alternative therapies are warranted. There is sufficient evidence to test the proof of concept that pathways targeted by statins will have a therapeutic effect in sarcoidosis, since, in pre-clinical studies, statins blunt Th1-mediated inflammatory responses.

Aims

The study involves a double-blind placebo-controlled, randomized trial which aims to determine if atorvastatin administration results in less steroid use and longer steroid-free intervals in patients with pulmonary sarcoidosis who require prednisone treatment.

Methods

Patients, who are 18-70 years old, with stage II or III pulmonary sarcoidosis, diagnosed by a compatible clinical history and supported by a lung, lymph node, or tissue biopsy, will be enrolled in the study, if they require prednisone therapy. The patients will be randomly assigned to two groups; as prednisone is tapered, one group will receive placebo and the other, atorvastatin. The two study drugs will be administered for twelve months, during which time patients will be periodically evaluated as to their clinical status and prednisone requirements. Pill counts and patient diaries will be used to determine the amount of steroid use during the study period. Patients with pulmonary fibrosis greater than 50 percent of total lung volume or severe co-morbidities will be excluded from the trial.

The primary endpoint is the duration of the steroid-sparing period. Secondary clinical and physiological endpoints are intended to analyze possible anti-inflammatory and beneficial effects of the drugs. Since there is no gold standard outcome measure in sarcoidosis, four categories of secondary endpoints will be used to characterize the effects of the therapeutic agent on the clinical course of the disease: imaging (high resolution chest CT); quality of life assessments (SF-36, and SGRQ), anti-inflammatory effects (biomarkers and relapse rates), and functional effects (CPET, PFTs). Finally, we will study the utility of exhaled nitric oxide and carbon monoxide in monitoring disease activity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients are eligible for the trial if they are 18-70 years old with radiographic stages II and III pulmonary sarcoidosis, and are on prednisone, methotrexate, or azathioprine for pulmonary sarcoidosis or who are steroid-requiring. Patients with extra-pulmonary sarcoidosis (except cardiac and neurosarcoidosis) may be eligible as long as they have active pulmonary (stage II or III) sarcoidosis.

Steroid-Requiring History:

A steroid-requiring patient is one who was previously stable but who ultimately experiences (a) increased symptoms associated with radiographic deterioration, and/or, (b) met the criteria for relapse and/or functional deterioration. In addition, patients who were prescribed prednisone for sarcoidosis, but have self-discontinued it (yet still have clinical and symptomatic disease and/or evidence of pulmonary functional deterioration) will be considered steroid-requiring.

This latter group of steroid-requiring patients is eligible for enrollment if they are willing to resume taking their latest stabilizing dose of prednisone for at least four weeks prior to study entry. If their dose cannot be determined, then 40 mg will be used.

Therefore, a history of symptomatic or clinical deterioration leading to therapy initiation, or a history of decline associated with attempts to decrease therapy should be established. Medical records review and discussion with the prescribing physician will be used to establish this history.

Radiographic Stages of Pulmonary Sarcoidosis:

STAGE< TAB> DESCRIPTION

0< TAB> Normal Chest Radiograph

I< TAB> Bilateral Hilar Lymphadenopathy

II< TAB> Pulmonary Infiltration and Bilateral Hilar Lymphadenopathy

III< TAB> Pulmonary Infiltration alone

Steroid-requiring refers to one of three situations:

Patients who meet relapse criteria or functional deterioration.

Functional deterioration criteria that warrants prednisone therapy includes:

If VC fell to 75% of the best recorded value for the patient before any treatment

If VC fell to greater than 50% of predicted value

IF DLCO fell to less than 60% of the best recorded value prior to their treatment

Patients who are on a previously prescribed systemic steroid, or alternative agent such as methotrexate or azathioprine, primarily for pulmonary sarcoidosis. Alternative agents must first be changed to roughly equivalent anti-inflammatory dose of prednisone and the patient should be stable on this dose for at least four weeks prior to randomization.

Patients who have substantial respiratory symptoms (distressing cough or dyspnea, which interferes with daily activities that would warrant therapy as per the standard of practice in the US.

Extra Pulmonary Sarcoidosis:

Patients with extra pulmonary sarcoidosis (except neurosarcoidosis and cardiac sarcoidosis) may be eligible as long as they have active pulmonary (stage II or III) sarcoidosis. All patients will be referred to an NIH ophthalmologist. Steroid therapy may be modified based upon the recommendations of the consultants, as well as per the lapse criteria described above.

EXCLUSION CRITERIA:

* Moderate to severe pulmonary fibrosis (stage IV sarcoidosis greater than 50% fibrosis)
* Lung Disease such as asthma, COPD, ILD (other than sarcoid-related)
* History of significant beryllium or asbestos exposure
* Pregnancy; or Active lactation/ child-bearing age female without appropriate birth control methods
* HIV disease
* Hepatitis C and Active Hepatitis B
* Other intervention protocols
* Immunosuppressive therapy (systemic or inhaled) other than corticosteroids or methotrexate
* Significant cardiac disease (NYSHA class greater than III), or serious coronary disease (unstable angina)
* Use of statins within 12 weeks of enrollment
* Allergies or intolerance to statins
* Liver disease (transaminases greater than 1.5X upper limits of normal) or cirrhosis
* Bleeding diathesis that is not correctable
* Inability to perform CPET (cycle ergometer) or PFT maneuvers
* Inability to understand the risks of the trial and the inability to complete the questionnaire
* Malignancy-- requiring chemotherapy or radiation therapy; except certain types of skin cancer that have been excised and have not spread.
* Myopathy, diagnosed via muscle biopsy (other than sarcoid-related myopathy); CPK grater than 1.5 upper limits of normal
* Surgical Risk Category [American Society of Anesthesiologists (ASA) class IV
* Ingestion of grapefruit juice or certain herbal preparations (see below), or medications that are potent inhibitors or inducers of the CYP3A4 system (see section 12.4 under precautions)
* Alcohol abuse (greater than 4 drinks/day)
* Bleeding into the brain or parts of the eyes (retina) (within the past year prior to enrollment)
* Uncontrolled Hypertension (SBP greater than 185 or DBP greater than 100 on two or more visits or assessments)
* Uncontrolled Diabetes Mellitus (Serum glucose level on two or more tests per day greater than 250 mg/dl or erratic blood sugar levels, noted on at least 2 or more assessments; and/or HgbA1C greater than 2x the upper limits of normal).
* Neurosarcoidosis
* Sarcoid Uveitis (Posterior Uveitis) or any Uveitis that cannot be managed with topical steroids alone, as determined by an ophthalmologist
* (Clinically apparent) Cardiac Sarcoidosis
* Active Smoker (Smoked within the past 2 months prior to randomization)
* Sickle cell disease (SS, SC, and sickle cell-beta thalassemia)
* Aseptic necrosis of the hip joints

Patients taking the following preparations will not be allowed to participate in the study unless they agree to discontinue usage at least two weeks prior to randomization and for the duration of the study period: grapefruit juice and herbal remedies that may lead to severe liver injury and/or muscle injury if taken with atorvastatin, including: Skullcap, chaparral, Germander, Jin Bu Huan, Valerian, Comfrey, and Eucalyptus. Since other products such as St. John s Wort, oat bran, and pectin can reduce the effectiveness of atorvastatin, they and similar agents, should also be discontinued at least two weeks before randomization and for the duration of the study period.

Subjects with inactive hepatitis B will require antiviral prophylaxis with an agent such as lamivudine, while on prednisone therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Fontana, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Statement on sarcoidosis. Joint Statement of the American Thoracic Society (ATS), the European Respiratory Society (ERS) and the World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) adopted by the ATS Board of Directors and by the ERS Executive Committee, February 1999. Am J Respir Crit Care Med. 1999 Aug;160(2):736-55. doi: 10.1164/ajrccm.160.2.ats4-99. No abstract available. PMID 10430755
- [Background] Newman LS, Rose CS, Maier LA. Sarcoidosis. N Engl J Med. 1997 Apr 24;336(17):1224-34. doi: 10.1056/NEJM199704243361706. No abstract available. PMID 9110911
- [Background] Thomas KW, Hunninghake GW. Sarcoidosis. JAMA. 2003 Jun 25;289(24):3300-3. doi: 10.1001/jama.289.24.3300. No abstract available. PMID 12824213
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0072.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by national advertising (self-referrals), physician referrals, and through a medical clinic sponsored by the NIH, from March 2006 through March 2015.
Pre-assignment Details: Subjects were screened by telephone and later during clinical testing a evaluation at the NIH Clinical Center. During this time subjects were evaluated to determine if they met the enrollment criteria, including that of treatment requiring disease, and relatively stable dosing prior to entry.
Groups:
- Intervention Group (Atorvastatin): Atorvastatin Subjects were assigned to the treatment intervention by way of double blind masking. Atorvastatin 80 mg/day was the initial treatment given, as tolerated for a 12 month period. During the study, a 50% dose reduction was applied for subjects meeting pre-specified criteria.
- Control Group (Placebo): Placebo In a double-blind fashion, subjects were assigned to receive the sham intervention which appeared the same as the intervention agent. For subjects meeting pre-specified criteria, a 50% dose reduction was applied during the 12 month treatment phase of the study.
Period: Overall Study
Arm/Group | Intervention Group (Atorvastatin) | Control Group (Placebo)
Started | 27 ("Started" meaning randomized) | 28
Completed | 24 | 24
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group (Atorvastatin): Atorvastatin: Subjects were assigned to the treatment intervention by way of double blind masking. Atorvastatin 80 mg/day was the initial treatment given, as tolerated for a 12 month period. During the study, a 50% dose reduction was applied for subjects meeting pre-specified criteria.
- Control Group (Placebo): Placebo: In a double-blind fashion, subjects were assigned to receive the sham intervention which appeared the same as the intervention agent. For subjects meeting pre-specified criteria, a 50% dose reduction was applied during the 12 month treatment phase of the study.
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Atorvastatin) | Control Group (Placebo) | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (7.95) | 46.8 (9.12) | 47.8 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: The Steroid Sparing Period
Description: The duration of steroid sparing was defined as the date when the target dose of prednisone was reached until the date at which the dose was increased and/or met the relapse (flare) criteria; or until the 12 month study phase ended if no prednisone dose increase was required. The steroid sparing period was measured in units of days. The prednisone target dose was defined as a 90% reduction of the baseline dose or an absolute prednisone dose of 4 mg/day or less.
Time Frame: 1 year
Measure: Mean (Inter-Quartile Range); unit: days
Groups:
- Control Group (Placebo): Placebo: In a double-blind fashion, subjects were assigned to receive the sham intervention which appeared the same as the intervention agent. For subjects meeting pre-specified criteria, a 50% dose reduction was applied during the 12 month treatment phase of the study: Placebo vs. Atorvastatin
Arm/Group | Intervention Group (Atorvastatin) | Control Group (Placebo)
Number analyzed (Participants) | 27 | 28
days | 301 [2 to 315] | 257 [152 to 322]

2. Secondary Outcome: Pulmonary Sarcoidosis Flares
Description: Flare rates and relative risk: Flares (relapses) were defined as the physiological deterioration in pulmonary function due to worsened pulmonary inflammation. The criteria used for a pulmonary flare included: > 15% decline in static function (FEV1 post, FVC post); or (> 20% DLCO adj); or a > 15% decline in walk distance as measured by the six minute walk test, or via a decline in oxygen consumption collected during a cardiopulmonary exercise test (CPET). Additional factors considered included an increase in dyspnea (>15% increase in the dyspnea scale (TDI); and/or significant radiographic worsening. Clinical assessment of the patient's status may have been factored into the criteria for flare determination as well.
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2017-09

3. Secondary Outcome: Pulmonary Function Tests
Description: Spirometry measurements (FVC and FEV1) obtained post-bronchodilator Diffusion, adjusted for hemoglobin
Time Frame: 12 month treatment period
Reporting Status: Not Posted, anticipated posting 2017-09

4. Secondary Outcome: Exercise Performance
Description: Cardiopulmonary Exercise Tests (VO2 peak, VO2/work, VECO2) Six minute Walk Test (distance, Borg scale)
Time Frame: 12 month treatment period
Reporting Status: Not Posted, anticipated posting 2017-09

5. Secondary Outcome: Quality of Life and Dyspnea Scales
Description: St. George's Respiratory Questionnaire SF-36 Modified MRC Dyspnea Scale
Time Frame: 12 month treatment period
Reporting Status: Not Posted, anticipated posting 2017-09

6. Other Pre Specified Outcome: Chest Imaging
Description: HRCT Chest radiographs
Time Frame: 12 month treatment period
Reporting Status: Not Posted, anticipated posting 2018-09

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention Group (Atorvastatin) | Control Group (Placebo)
Serious Adverse Events (participants affected / at risk) | 12/27 | 16/28
Other Adverse Events (participants affected / at risk) | 16/27 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (Atorvastatin) (N=27) | Control Group (Placebo) (N=28)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate Aminotransferase elevation (Hepatobiliary disorders) | 1 (1) | 1 (1)
Alanine aminotransferase elevation (Investigations) | 1 (1) | 0 (0)
Aldolase increased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Creatinine Phosphokinase Increase (Investigations) | 0 (0) | 1 (1)
Deep Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Diffusion of carbon monoxide (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Myoglobin Increase (Investigations) | 0 (0) | 1 (1) — Rhabdomyolysis
Obstructive Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Temperature Elevation (Infections and infestations) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Muscle Weakness unilateral (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (Atorvastatin) (N=27) | Control Group (Placebo) (N=28)
Aldolase Increase (Investigations) | 2 (2) | 3 (3)
ACE Level increased (Investigations) | 2 (2) | 1 (1)
Alkaline Phosphatase Increase (Investigations) | 3 (3) | 1 (1)
Alanine aminotransferase Increased (Investigations) | 13 (13) | 4 (4)
Asparatate aminotransferase Increased (Investigations) | 14 (14) | 5 (5)
Amylase Increased (Investigations) | 0 (0) | 4 (4)
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Creatine Phosphokinase increased (Investigations) | 2 (2) | 3 (3)
Creatinine increased (Investigations) | 0 (0) | 4 (4)
Diffusion of Carbon Monoxide decreased (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Lipase Increase (Investigations) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The recruitment goal of 96 subjects was not met due to slow accrual. The primary endpoint analysis was based on the available subject data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No